CLINICAL TRIAL: NCT04950075
Title: A Randomized, Blinded, Placebo-controlled, Phase 2 Study of INBRX-109 in Unresectable or Metastatic Conventional Chondrosarcoma
Brief Title: Study of INBRX-109 in Conventional Chondrosarcoma
Acronym: ChonDRAgon
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Inhibrx Biosciences, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Ph2 INBRX-109 SA CS
Record Dates: First submitted 2021-06-14; First posted 2021-07-06 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Conventional Chondrosarcoma
Keywords: DR5; INBRX-109; Apoptosis; Programmed cell death

STUDY DESIGN:
Intervention Model Description: INBRX-109 and placebo arms are in parallel. Patients on placebo are allowed to cross-over to open-label INBRX-109 at time of disease progression.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- INBRX-109 (Experimental): IV every three weeks
  Interventions: Drug: INBRX-109
- Placebo (Placebo Comparator): IV every three weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: INBRX-109 — Tetravalent DR5 Agonist Antibody
  Arms: INBRX-109
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
Randomized, blinded, placebo-controlled, Phase 2 study of INBRX-109 in unresectable or metastatic conventional chondrosarcoma patients.

DETAILED DESCRIPTION:
This is a randomized, blinded, placebo-controlled, Phase 2 study of INBRX-109 in unresectable or metastatic conventional chondrosarcoma patients. INBRX-109 is a recombinant humanized tetravalent antibody targeting the human death receptor 5 (DR5).

ELIGIBILITY:
Inclusion Criteria:

1. Conventional chondrosarcoma, unresectable (=inoperable) or metastatic.
2. Measurable disease by RECISTv1.1. Note: Tumor lesions located in a previously irradiated (or other locally treated) area will be considered measurable, provided there has been clear imaging-based progression of the lesions since the time of treatment.
3. Radiologic progression of disease per RECISTv1.1 criteria within 6 months prior to screening for this study.
4. Adequate hematologic, coagulation, hepatic and renal function as defined per protocol.
5. Eastern Cooperative Oncology Group performance status (ECOG PS) of 0 or 1.
6. Estimated life expectancy of at least 12 weeks.
7. Availability of archival tissue or fresh cancer biopsy are mandatory.

Exclusion Criteria:

1. Any prior exposure to DR5 agonists.
2. Allergy or sensitivity to INBRX-109 or known allergies to CHO-produced antibodies.
3. Non-conventional chondrosarcoma, e.g., clear-cell, mesenchymal, extraskeletal myxoid, myxoid, and dedifferentiated chondrosarcoma.
4. Prior or concurrent malignancies. Exception: Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessments.
5. Chronic liver diseases. Exception: Patients with fatty liver disease are acceptable as long as adequate hepatic function as defined in the inclusion/exclusion criteria is confirmed.
6. Evidence or history of multiple sclerosis (MS) or other demyelinating disorders.
7. Other exclusion criteria per protocol.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 206 (Actual)
Dates: Start 2021-09-23 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival per RECISTv1.1 by real time IRR comparing INBRX-109 and placebo | 3 years
  Progression-free survival per RECISTv1.1 will be determined.

SECONDARY OUTCOMES:
Overall survival of patients comparing INBRX-109 and placebo | 3 years
  Overall Survival in the ITT population
ORR per RECISTv1.1 by real-time IRR. | 3 years
  Tumor response will be determined by RECISTv1.1.
PFS per RECISTv1.1 by Investigator assessment | 3 years
  PFS per RECISTv1.1, by Investigator assessment, comparing INBRX-109 and placebo.
Quality of life assessed by EORTC questionnaire for cancer patients (QLQ-C30) comparing INBRX-109 and placebo | 3 years
  Quality of life will be determined.
DCR per RECISTv1.1 by real-time IRR | 3 years
  measured by DCR per RECISTv1.1, assessed by central real-time IRR, comparing INBRX-109 and placebo
DOR per RECISTv1.1 by real-time IRR | 3 years
  evaluate duration of response (DOR) per RECISTv1.1, assessed by central real-time IRR, comparing INBRX-109 and placebo
To evaluate the safety and tolerability of INBRX-109 | 3 years
  Adverse events will be assessed and severity assigned by using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 5.0.
Characterize the pharmacokinetics of INBRX-109. | 3 years
  AUC0-inf, AUC0-last, AUC0-21d, Cmax, Ctrough, Tmax will be estimated using a standard non-compartmental method as the data allow. Other PK parameters (λz, t½, Vd, CL, and accumulation ratios RCmax, RCtrough) will be calculated if data permit.
Immunogenicity of INBRX-109 | 3 years
  Frequency of anti-drug antibodies against INBRX-109 will be determined.

OTHER OUTCOMES:
Evaluate Quality of Life | 3 years
  QoL per EORTC QLQ-C30, EQ-5D-5L, PGI-C, PGI-S
Potential predictive response biomarkers | 3 years
  Evaluate the relationship between potential predictive response biomarkers and efficacy of INBRX-109
PFS per RECISTv1.1 by Investigator assessment | 3 years
  evaluate the anticancer efficacy of INBRX-109 as measured by PFS (by Investigator assessment) for crossover population after treatment with INBRX-109
ORR per RECISTv1.1 by Investigator assessment | 3 years
  evaluate the anticancer efficacy of INBRX-109 as measured by ORR (by Investigator assessment) for crossover population after treatment with INBRX-109

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Lead, Study Director — Inhibrx Biosciences, Inc
Locations (68):
- United States (32):
  - Mayo Clinic Cancer Center, Phoenix, Arizona
  - Precision NextGen Oncology & Research Center, Beverly Hills, California
  - University of California, San Francisco (UCSF), San Francisco, California
  - Sarcoma Oncology Center, Santa Monica, California
  - University of Colorado, Denver, Colorado
  - Yale Cancer Center, New Haven, Connecticut
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Northwestern University - Robert H. Lurie Comprehensive Cancer Center, Chicago, Illinois
  - Rush Cancer Center, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - Johns Hopkins, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Washington University School of Medicine - St. Louis, St Louis, Missouri
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Columbia University, New York, New York
  - Duke University, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - University of Oklahoma - Stephenson Cancer Center, Oklahoma City, Oklahoma
  - Oregon Health & Science University (OHSU) Knight Cancer Institute, Portland, Oregon
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Texas Southwestern, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia
  - University of Washington, Seattle, Washington
- Australia (3):
  - Royal Adelaide Hospital, Adelaide
  - Chris O'Brien Lifehouse, Camperdown
  - Princess Alexandra Hospital, Woolloongabba
- France (9):
  - Institut Bergonie, Bordeaux, Cedex
  - Centre Oscar Lambret, Lille
  - Centre Leon Berard, Lyon
  - AP-HM - Hôpital de la Timone, Marseille
  - ICM - Institut Regional du Cancer de Montpellier, Montpellier
  - Centre Antoine-Lacassagne, Nice
  - AP-HP Hopital Cochin, Paris
  - Centre Eugene Marquis, Rennes
  - Gustave Roussy, Villejuif
- Germany (4):
  - Helios Klinikum Berlin-Buch, Berlin
  - Universitaetsklinikum Heidelberg, Heidelberg
  - Universitätsmedizin Mannheim, Mannheim
  - Universitaetsklinikum Tuebingen, Tübingen
- Saint Vincent's University Hospital part of Irish Sarcoma Group, Dublin, Ireland
- Italy (6):
  - IRCCS Istituto Ortopedico Rizzoli di Bologna, Bologna
  - La Fondazione e l'Istituto di Candiolo, Candiolo
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone, Palermo
  - Nuovo Ospedale di Prato, Prato
  - Policlinico Universitario Campus Biomedico, Roma
- Netherlands (2):
  - Groningen UMC, Groningen
  - Leiden University Medical Center, Leiden
- Spain (7):
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital de la Santa Creu i Sant Pau Barcelona, Barcelona
  - Hospital Clinico San Carlos, Madrid
  - Hospital Fundación Jiménez Díaz, Madrid
  - Hospital Clinico Universitario de Santiago, Santiago de Compostela
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Universitari i Politecnic La Fe, Valencia
- United Kingdom (4):
  - University College London Hospital (UCL), London
  - Royal Marsden NHS Foundation Trust, London
  - The Christie NHS Foundation Trust, Manchester
  - Churchill Hospital, Oxford

IPD SHARING:
Plan to Share IPD: No